CLINICAL TRIAL: NCT02363920
Title: Short Term Physiological Effects of Nasal High Oxygen Flow vs Low Oxygen Flow and Noninvasive Ventilation (NIV) on Respiratory Mechanics
Brief Title: Short Term Physiological Effects of Nasal High Flow Oxygen on Respiratory Mechanics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief of Respiratory and Critical care Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 402015
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: COPD; Chronic Hypercapnic Respiratory Failure
Keywords: COPD patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- spontaneous breathing trial (Placebo Comparator): the patients will be asked to breathe spontaneously using their acutal low oxygen flow
  Interventions: Device: HOF; Device: noninvasive mechanical ventilation (NIV)
- HOF20 (Active Comparator): the patients will be asked to breathe with HOF of 20 L/min
  Interventions: Device: HOF; Device: noninvasive mechanical ventilation (NIV)
- HOF30 (Active Comparator): the patients will be asked to breathe with HOF of 30 L/min
  Interventions: Device: HOF; Device: noninvasive mechanical ventilation (NIV)
- noninvasive mechanical ventilation (NIV) (Active Comparator): the patients will be asked to breathe with the support of a ventilator via a oro-nasal interface
  Interventions: Device: HOF; Device: noninvasive mechanical ventilation (NIV)

INTERVENTIONS:
Device: HOF — the addition of high oxygen flow to patients breathing spontaneously
Device: noninvasive mechanical ventilation (NIV) — the addition of a ventilatory support delivered with a oro-nasal interface

SUMMARY:
Nasal High Oxygen Flow (HOF) has been demonstrated to reduce the re-intubation rate in hypoxic patients and ameliorate breathing pattern in hypercapnic patients.

The aim of this study is to better understand the physiological mechanism underlying these results, assessing the respiratory mechanics in stable hypercapnic COPD patients.

DETAILED DESCRIPTION:
Subjects. 10 in-patients with stable COPD and chronic hypercapnic respiratory failure with no history of neurological or chronic cardiac disease will be recruited. They need to be in a phase of clinical stability and were for a short period of rehabilitation. Patients with X-ray evidence of pulmonary edema or congestion and pulmonary infiltrate will be excluded from the study. Written consent will be obtained from all subjects, and the protocol will be approved by the Ethics Committee.

Measurements. Static and dynamic lung volumes assessed by body plethysmography (MasterLab-Jaeger, Hochberg, Germany).

Flow measured with a pneumotachograph (Screenmate Box 0586, Jaeger GmbH, Hochberg, Germany), connected to a rigid mouthpiece.

Airway pressure measured through tubing inserted in the mouthpiece and connected to a differential pressure transducer (Honeywell 300 cm H2O, Freeport, IL, USA). VT obtained by integration of the flow signal. The inspiratory (TI), expiratory (TE) and total breathing cycle (TTOT) duration, respiratory frequency (RR), and duty cycle (TI/TTOT) calculated as average values of 10 consecutive breaths, after 5 minutes of breathing.

Baseline from peak changes in esophageal (Pes), gastric (Pga), and transdiaphragmatic (Pdi) pressures measured using the balloon-catheter technique. Pressure at the airway opening (Paw) measured via a side port.

Respiratory mechanics will be assessed using Mead and Wittenberger's technique. Inspiratory pulmonary resistance (R,L) and elastance (E,L) calculated by fitting the equation of motion of a single-compartment model using multilinear regression.

Dynamic PEEPi (PEEPi,dyn) will be measured according to Appendini et al. The pressure time integrals of the diaphragm and the other inspiratory muscles calculated per breath (PTPdi/b and PTPes/b, respectively) and per minute (PTPdi/min and PTPes/min).

Subjective ratings of dyspnea assessed during the various trials using Borg's scale.

Arterial blood gases (ABGs) measured in samples taken from the radial artery (ABL 550 Radiometer, Copenhagen, Denmark).

The above mentioned variables, excluding arterial blood gases recorded after 15 minutes of spontaneous breathing. At the end of this part of the study, the patients will undergo a randomized 30' trial of: 1) non-invasive mechanical ventilation (NIMV) through a nose mask for 20 minutes while they were in a sitting position. The following pressures will be used: 14 cmH2O of inspiratory aid and 4 cmH2O of expiratory-positive airway pressure. 2) HOF at the flow of 20 L/min 3) HOF at the flow of 30 L/min ECG, SaO2 will be continuosly recorded All signals collected using a personal computer equipped with an A/D board, and stored at a sampling rate of 100 Hz. The mean value of each physiological variable during the 5 minutes of recording used for analyses. Results presented as mean + standard deviation (SD). Differences between physiological parameters recorded in the 3 settings will be analysed by paired Student's T-test. Pearson's coefficient will be used to calculate to assess correlation between variables. A p value <0.05 chosen as the threshold of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Chronic hypercapnic respiratory failure (pH>7.34 and PaCO2>45 mmHg)

Exclusion Criteria:

* Cancer
* Neurological and cardiac disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
recording of respiratory mechanics | 30 minutes per arm
  Respiratory mechanics will be assessed using Mead and Wittenberger's technique.

SECONDARY OUTCOMES:
dyspnea score | 30 minutes per arm
  dyspnea will be recorded using the Borg scale that is a numeric scale where 0 is no dyspnea and 10 the maximal dyspnea that a patient can imagine

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, md, Principal Investigator — Sant'Orsola Malpighi Hospital
Locations (1):
- San'Orsola Malpighi Hospital, Bologna ITALY, Bologna, Italy

REFERENCES:
- [Derived] Pisani L, Fasano L, Corcione N, Comellini V, Musti MA, Brandao M, Bottone D, Calderini E, Navalesi P, Nava S. Change in pulmonary mechanics and the effect on breathing pattern of high flow oxygen therapy in stable hypercapnic COPD. Thorax. 2017 Apr;72(4):373-375. doi: 10.1136/thoraxjnl-2016-209673. Epub 2017 Jan 19. PMID 28104830